CLINICAL TRIAL: NCT03107130
Title: Complex Urodynamic Testing: Who Requires it? A Retrospective Review
Brief Title: Urodynamic Studies Prior to Surgery for Stress Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 17-004
Record Dates: First submitted 2017-03-14; First posted 2017-04-11 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Urodynamic Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SUI Surgery Patients in 2015: All women 18 years of age or older, who underwent surgery for SUI between January 2015 and December 2015

SUMMARY:
This retrospective descriptive study is to determine what proportion of Cincinnati Urogynecology Associates patients who underwent surgical management for stress urinary incontinence (SUI) would qualify for a basic office exam (BOE) alone, using the inclusion and exclusion criteria of the Value of Urodynamic Evaluation (VALUE) trial, and thus could have potentially had Urodynamic studies (UDS) omitted from their preoperative workup.

DETAILED DESCRIPTION:
Urodynamic studies (UDS) are an assessment tool used to evaluate physiologic variables during bladder filling, bladder storage, and bladder emptying. They are commonly performed as part of the routine preoperative evaluation of women with symptoms of SUI. However, UDS are costly, with payments allowed by Medicare quoted at greater than $500, time consuming, uncomfortable, and have been shown to increase the risk of urinary tract infection. But most concerning is the fact that UDS have not been shown to improve surgical outcomes.

In 2012, the Value of Urodynamic Evaluation (VALUE) trial evaluated 630 women who underwent a basic office exam (BOE) or BOE plus UDS, and concluded that for women with uncomplicated, demonstrable SUI a BOE alone was not inferior to evaluation with UDS for outcomes at 1 year. This recent publication has resulted in urogynecology practices across the country evaluating their own standard of care when it comes to preoperative evaluation of SUI.

Cincinnati Urogynecology Associates, TriHealth Inc. standard practice is to perform UDS on all patients undergoing surgery for SUI. The providers of Cincinnati Urogynecology Associates, TriHealth Inc. would be remiss if the providers did not follow this trend and evaluate their own personal practice of preoperative UDS in patients presenting with SUI.

ELIGIBILITY:
Inclusion Criteria:

* All women 18 years of age or older
* Underwent surgery for SUI performed by a physician at Cincinnati Urogynecology Associates, TriHealth Inc. between January 2015 and December 2015

Exclusion Criteria:

* Age < 18 years old
* Concomitant surgery for anterior or apical pelvic organ prolapse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women 18 years of age or older, who under went surgery for SUI performed by a physician at Cincinnati Urogynecology Associates, TriHealth Inc. between January 2015 and December 2015
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who meet VALUE trial criteria | Within 15 months to the initial presentation
  A patient meets all the inclusion criteria and doesn't meet any of exclusion criteria of the VALUE trial will be classified under the category of who meets VALUE trial criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nager CW, Brubaker L, Litman HJ, Zyczynski HM, Varner RE, Amundsen C, Sirls LT, Norton PA, Arisco AM, Chai TC, Zimmern P, Barber MD, Dandreo KJ, Menefee SA, Kenton K, Lowder J, Richter HE, Khandwala S, Nygaard I, Kraus SR, Johnson HW, Lemack GE, Mihova M, Albo ME, Mueller E, Sutkin G, Wilson TS, Hsu Y, Rozanski TA, Rickey LM, Rahn D, Tennstedt S, Kusek JW, Gormley EA; Urinary Incontinence Treatment Network. A randomized trial of urodynamic testing before stress-incontinence surgery. N Engl J Med. 2012 May 24;366(21):1987-97. doi: 10.1056/NEJMoa1113595. Epub 2012 May 2. PMID 22551104